CLINICAL TRIAL: NCT00785915
Title: A Phase I, Single-center, Randomized, Double-blind, Placebo-controlled Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD6765 in Healthy Male and Female Japanese and Caucasian Subjects
Brief Title: AZD6765 Single and Multiple Ascending Dose Study in Healthy Male and Female Japanese and Caucasian Subjects
Acronym: JSAD/JMAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6702C00013
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: AZD6765; Japanese and Caucasian Healthy Volunteers; Phase I study; Single and multiple Ascending Dose; Japanese volunteers
MeSH Terms: interventions — AZD6765

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD6765
- 2 (Placebo Comparator): given (2 subjects in each ethnic/dose group)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6765 — single administration and once daily for 5 days
  Arms: 1
Drug: Placebo — single administration and once daily for 5 days
  Arms: 2

SUMMARY:
This is a Phase I randomized double-blind, placebo-controlled, single and multiple ascending dose study to assess the safety, tolerability and pharmacokinetics of AZD6765 in healthy male and female Japanese and Caucasian subjects

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI): 18 to 27 kg/m 2
* Female subjects must be postmenopausal for at least 1 year, surgically sterile, or using a reliable method of contraception at screening.
* Male subjects must be willing to use accepted contraceptive methods, avoid unprotected sex, and donating sperm until 3 months after drug administration.

Exclusion Criteria:

* Clinically relevant disease and/or abnormalities (past or present)
* Clinically relevant abnormalities in physical examinations,vital signs,clinical chemistry, hematology or urinalysis at screening as judged by the investigator
* Use of any prescription medication within 14 days of Day 1
* Use of over-the-counter (OTC) medication (with the exception of acetaminophen), vitamin/nutritional supplements and herbal preparations within 14 days of Day 1
* Smoking in excess of 5 cigarettes per day or the equivalent within 28 days of Day 1

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability; Adverse events (AEs), vital signs, physical examinations, ECGs and clinical laboratory assessments | During the study

SECONDARY OUTCOMES:
Pharmacokinetic - Pharmacokinetic parameters for AZD6765 in plasma and urine | During residential period
Genetics; Collect blood samples for optional exploratory genetic studies focusing on identification of genes that influence the disposition, efficacy, safety and tolerability of AZD6765. | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yen, MD, Principal Investigator — California Clinical Trials
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Baltimore, Maryland

REFERENCES:
- See also: D6702C00013 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=573&filename=D6702C00013_Clinical_Study_Report_Synopsis.pdf